CLINICAL TRIAL: NCT00866892
Title: A Pilot Study of Noncontaminated Facial and Scalp Wounds in the Pediatric Population: Getting Away Without Irrigation and Scrubbing
Brief Title: Pediatric Pilot Study: Irrigation and Scrubbing in Facial and Scalp Wounds
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Jeffrey Louie, MD, Children's Hospitals and Clinics of Minnesota
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0808-081
Record Dates: First submitted 2009-03-19; First posted 2009-03-23 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Facial and Scalp Lacerations
MeSH Terms: conditions — Facies | interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- irrigation (Active Comparator)
  Interventions: Procedure: Irrigation
- no irrigation (Experimental)
  Interventions: Procedure: No irrigation

INTERVENTIONS:
Procedure: Irrigation — irrigation
  Arms: irrigation
Procedure: No irrigation — no irrigation
  Arms: no irrigation

SUMMARY:
Most pediatric lacerations occur indoors and are considerably noncontaminated. Wounds that occur outside of the house where dirt often enters the laceration, irrigation and scrubbing with soap has been proven effective at decreasing post-laceration infections. To date there are no pediatric prospective studies addressing a less aggressive approach to face and scalp wound preparation in pediatrics. We argue that wiping wounds with sterile gauze soaked in sterile saline will not increase infection rates as compared to our current practice. In our emergency departments, the current standard of care for all lacerations is aggressive wound preparation: irrigation and scrubbing. This occurs regardless if the wound is contaminated or not. Research has proven that irrigation and scrubbing is unwarranted in adults with face and scalp lacerations. We want to perform a pilot/feasibility study comparing our two emergency campuses. One campus will serve as the control site, while the other will be the intervention site. In this pilot study, our goal is to demonstrate the feasibility of the intervention and provide data that a less aggressive approach to wound preparation is just as effective as our standard of care. We hope this project leads to further discussion about how we manage noncontaminated lacerations and provides a stepping-stone to a larger, appropriated powered study.

ELIGIBILITY:
Inclusion Criteria:

1. facial and scalp wounds acquired by blunt trauma,
2. wounds incurring within a house or indoor gym,
3. all ages, 1 month to 20 years of age.

Scalp is defined as the skin covering the head. The face is the area anterior to the ears, below the chin and extending to the hairline of the forehead. Wounds requiring deep sutures will also be included.

Exclusion Criteria:

1. Patients presenting with wounds that occur outdoors,
2. Wounds greater than 12 hour old,
3. Immunocompromised, malnourished or a diabetic,
4. Intoxicated,
5. Currently on antibiotics,
6. Sickle cell anemia,
7. Collagen vascular disease,
8. Wounds requiring plastic surgery,
9. Wounds from human or animal bites,
10. Wounds not on the face or scalp,
11. Patient's just discharged from the hospital within 72 hours,
12. Wounds with foreign bodies or grossly contaminated,
13. No suture nurses are present or available to suture.

Ages: 1 Month to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Our specific aim is to provide evidence that using a less aggressive approach to wound preparation in a selective population will be as effective as our current practice. | 12 months

SECONDARY OUTCOMES:
Our secondary goals are to involve nurses in a prospective interventional study, document the feasibility of the study, and demonstrate patient satisfaction with our suture outcomes. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Louie, MD, Principal Investigator — Children's Hospitals and Clinics of Minnesota; Russell Grimsby, RN, Principal Investigator — Children's Hospitals and Clinics of Minnesota; Michael Oakes, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Saint Paul and Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Stussman BJ. National Hospital Ambulatory Medical Care Survey: 1994 emergency department summary. Adv Data. 1996 May 17;(275):1-20. No abstract available. PMID 10162000
- [Background] Hollander JE, Singer AJ, Valentine S, Henry MC. Wound registry: development and validation. Ann Emerg Med. 1995 May;25(5):675-85. doi: 10.1016/s0196-0644(95)70183-4. PMID 7741347
- [Background] Islam S, Ansell M, Mellor TK, Hoffman GR. A prospective study into the demographics and treatment of paediatric facial lacerations. Pediatr Surg Int. 2006 Oct;22(10):797-802. doi: 10.1007/s00383-006-1768-7. Epub 2006 Sep 1. PMID 16947027
- [Background] Baker MD, Lanuti M. The management and outcome of lacerations in urban children. Ann Emerg Med. 1990 Sep;19(9):1001-5. doi: 10.1016/s0196-0644(05)82563-6. PMID 2393165
- [Background] Sagerman PJ. Wounds. Pediatr Rev. 2005 Feb;26(2):43-9. doi: 10.1542/pir.26-2-43. No abstract available. PMID 15687474
- [Background] Krizek TJ, Davis JH. Endogenous wound infection. J Trauma. 1966 Mar;6(2):239-48. No abstract available. PMID 5908175
- [Background] Haury B, Rodeheaver G, Vensko J, Edgerton MT, Edlich RF. Debridement: an essential component of traumatic wound care. Am J Surg. 1978 Feb;135(2):238-42. doi: 10.1016/0002-9610(78)90108-3. PMID 626301
- [Background] Hollander JE, Singer AJ, Valentine S. Comparison of wound care practices in pediatric and adult lacerations repaired in the emergency department. Pediatr Emerg Care. 1998 Feb;14(1):15-8. doi: 10.1097/00006565-199802000-00004. PMID 9516624
- [Background] Valente JH, Forti RJ, Freundlich LF, Zandieh SO, Crain EF. Wound irrigation in children: saline solution or tap water? Ann Emerg Med. 2003 May;41(5):609-16. doi: 10.1067/mem.2003.137. PMID 12712026
- [Background] Hollander JE, Richman PB, Werblud M, Miller T, Huggler J, Singer AJ. Irrigation in facial and scalp lacerations: does it alter outcome? Ann Emerg Med. 1998 Jan;31(1):73-7. doi: 10.1016/s0196-0644(98)70284-7. PMID 9437345